CLINICAL TRIAL: NCT05484414
Title: A 2 Part Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Pharmacokinetics of SAD/MAD Oral Doses of SRP-3D (DA), and to Characterize the Effect of Food on the Pharmacokinetics in Healthy Male and Female Subjects
Brief Title: Safety and Pharmacokinetics of SAD/MAD Oral Doses of SRP-3D (DA)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: South Rampart Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRP-101
Record Dates: First submitted 2022-07-27; First posted 2022-08-02 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Pain
Keywords: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): SRP-3D (Diethylamide) Oral Suspension, 100 mg/mL
  Interventions: Drug: SRP-3D (diethylamide)
- Placebo (Placebo Comparator): Matching Placebo for SRP-3D (Diethylamide) Oral Suspension, 100 mg/mL
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SRP-3D (diethylamide) — SRP-3D (Diethylamide) Oral Suspension, 100 mg/mL
  Other Names: SRP-3D (DA)
  Arms: Experimental
Drug: Placebo — Matching Placebo for SRP-3D (Diethylamide) Oral Suspension, 100 mg/mL
  Other Names: Control
  Arms: Placebo

SUMMARY:
This is a two-part randomized, double-blind, placebo-controlled study.

DETAILED DESCRIPTION:
This is a two-part randomized, double-blind, placebo-controlled study. The study comprises a SAD (Part 1) assessment which will include a food effect assessment that contributes data to inform a subsequent MAD (Part 2) dose-ranging study. Safety measurements will be collected throughout the study for all subjects. Blood samples will be collected to determine the PK parameters of SRP-3D (DA).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female. Females must not be pregnant or breastfeeding.
2. Is between 18 and 55 years of age (inclusive).
3. Able to speak and understand English or Spanish.
4. Agrees to comply with testing procedures.
5. Has a body mass index (BMI) between 18.0 and 32.0 kg/m2 (inclusive).
6. The subject meets good health criteria.
7. Females of non-childbearing potential or agree to use birth control.
8. Male subjects must be surgically sterile or agree to the use birth control.
9. Agree to the confinement period and return for the outpatient visits.
10. Has vital signs at screening within appropriate ranges.

Exclusion Criteria:

1. History or presence of clinically significant diseases.
2. Abnormal diet 4 weeks preceding the first dose of study medication.
3. Received any investigational product in a clinical study.
4. Previously been administered IMP in this study.
5. Taking any prescribed or OTC drug.
6. Taking moderate or strong inhibitors/inducers of cytochrome P450.
7. History of hypersensitivity to acetaminophen or similar chemical entities.
8. Presence or history of allergy or blood or plasma donation.
9. Blood or plasma donation
10. Smokers and those who have smoked within the last 12 months.
11. Current users of e-cigarettes and nicotine replacement products.
12. Consumption of prohibited beverages or foods.
13. Prior history of substance abuse or treatment.
14. Regular alcohol consumption.
15. Positive alcohol urine test at screening or admission.
16. Is a female with a positive pregnancy test result.
17. Positive urine screen for drugs of abuse.
18. Positive test for hepititus B or C, or HIV.
19. Active infection, periodontal disease,. certain dental appliances.
20. Glucose-6-phosphate-dehydrogenase (G6PD) deficiency.
21. Significant serious skin disease.
22. Cohort 3 only: history of cholecystectomy or gall stones.
23. Have poor venous access that limits phlebotomy
24. Evidence of current SARS-CoV-2 infection
25. Clinically significant abnormal clinical chemistry, hematology or urinalysis.
26. Immediate family members of a study site or Sponsor employee.
27. Failure to satisfy the Investigator of fitness to participate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-07-16 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | The time of providing written informed consent until 30 days after the last dose of study drug
  Reported AEs

SECONDARY OUTCOMES:
PK parameters 1 | 6 days
  Lag time (Tlag)
PK parameters 2 | 6 days
  Time to reach maximum (peak) plasma concentration following drug administration (Tmax)
PK parameters 3 | 6 days
  Maximum (peak) plasma drug concentration (Cmax)
PK parameters 4 | 6 days
  Area under the plasma concentration-time curve from time zero to infinity (AUCinf)
PK parameters 5 | 6 days
  Area under the plasma concentration-time curve from time zero to infinity (AUClast)
PK parameters 6 | 6 days
  Area under the plasma concentration-time curve (AUC0-tau)
PK parameters 7 | 6 days
  Terminal disposition rate constant/terminal rate constant (λz)
PK parameters 8 | 6 days
  Elimination half-life (T1/2)
PK parameters 9 | 6 days
  Apparent total clearance of the drug from plasma after oral administration (CL/F)
PK parameters 10 | 6 days
  Apparent volume of distribution during terminal phase after non-intravenous administration (Vz/F)

CONTACTS AND LOCATIONS:
Overall Officials: Hernan A Bazan, MD, Study Chair — CEO
Locations (1):
- Quotient Sciences-Miami, Inc., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No